CLINICAL TRIAL: NCT01038791
Title: Patients-ventilator Interaction During Sleep: the Role of Humidification. A Pilot Short Term Study
Brief Title: Patients-ventilator Interaction During Sleep: Effect of Humidification System
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, dr. Stefano Nava, Chief ICU, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 593
Record Dates: First submitted 2009-12-16; First posted 2009-12-24 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2013-01

CONDITIONS: Chronic Hypercapnic Respiratory Failure
Keywords: chronic hypercapnic respiratory failure; COPD; RTD; sleep architecture; humidification
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- usual ventilation (Active Comparator): application of usual mechanical ventilation without humidification system
  Interventions: Device: usual mechanical ventilation without humidification
- heated humidifier (Experimental): mechanical ventilation with heated humidifier
  Interventions: Device: heated humidification
- heat and moisture exchanger (Experimental): mechanical ventilation with heat and moisture exchanger
  Interventions: Device: heat and moisture exchanger

INTERVENTIONS:
Device: heated humidification — temperature 35°
  Other Names: HH
  Arms: heated humidifier
Device: heat and moisture exchanger — single patient device
  Other Names: HME
  Arms: heat and moisture exchanger
Device: usual mechanical ventilation without humidification — mechanical ventilation with usual parameters
  Other Names: control
  Arms: usual ventilation

SUMMARY:
At present, little data is available in the medical literature regarding the affects of humidification on NIMV efficacy, sleep quality and upper airway symptoms in patients undergoing nocturnal NIMV.

The aim of the present pilot study is to assess the impact of two humidification systems on sleep quality, NIMV efficacy, patient-ventilator interaction, prevalence of NIMV side effects, compliance to treatment, in a group of stable patients already enrolled in a long-term nocturnal mechanical ventilation program for chronic hypercapnic respiratory failure or sleep hypoventilation.

DETAILED DESCRIPTION:
BACKGROUND Non-invasive mechanical ventilation (NIMV), usually delivered during night time, is widely used at home in chronic hypercapnic respiratory, both in patients with COPD and restrictive thoracic diseases (RTD). The aim of chronic NIMV is to improve daytime arterial blood gases, sleep quality decreasing symptoms of hypoventilation (mainly during sleep), quality of life and mood.

Scarce data is available about the NIMV compliance at home; poor compliance may reduce the positive effects of mechanical ventilation. Previous data shows that patients enrolled to long-term home ventilation program may drop out early, mainly because of skin irritation, upper airway problems, and air leaks.

Studies performed on patients with sleep apnea, receiving CPAP therapy at home, showed that the occurrence of leaks during ventilation can cause the development of mucosal inflammation, nasal congestion and increased nasal airways resistance. On the other hand, the presence or the development of nasal obstruction makes the arise or the worsening of air leaks (the vicious cycle) more reliable.

A lack of humidification may increase nasal resistance and nasal symptoms and, therefore, contribute to reduction in compliance. Furthermore, leaks may have significant consequences on inspiratory and expiratory trigger functions, inducing poor patient-ventilator interactions. Indeed, the presence of ineffective efforts, the most common phenomenon of bad patient-ventilation interactions, is very common in patients receiving long term home ventilation and usually associated with poorer gas exchange during sleep.

At present, little data is available in the medical literature regarding the affects of humidification on NIMV efficacy, sleep quality and upper airway symptoms in patients undergoing nocturnal NIMV.

The aim of the present pilot study is to assess the impact of two humidification systems on sleep quality, NIMV efficacy, patient-ventilator interaction, prevalence of NIMV side effects, compliance to treatment, in a group of stable patients already enrolled in a long-term nocturnal mechanical ventilation program for chronic hypercapnic respiratory failure or sleep hypoventilation.

PATIENTS We plan to enrol 20 patients with chronic respiratory failure or sleep hypoventilation already included in a long-term home non-invasive ventilation program (at least 3 months).

Inclusion criteria Patients in stable conditions (no acute exacerbations in the 4 weeks before enrolment), well adapted to ventilation and without problems with the ventilation mask.

Exclusions criteria Patients with acute respiratory failure, recent exacerbations, severe co-morbidities (i.e. hearth failure, recent stroke etc.) Recent upper airways surgery. Allergic rhinitis, severe nasal stenosis.

STUDY DESIGN

Patients will undergo three consecutive nocturnal polysomnographs. Patients will have a baseline therapy of NIMV without humidification for 1 week. They will then undergo a nocturnal polysomnograph on the last evening of the baseline therapy. Patients will then be randomly assigned to use HH or HME for 1 week and undergo a nocturnal polysomnography on the last evening . The patients will then be assigned to the second method of humidification for 1 week and undergo a third nocturnal polysomnograph on the last evening. The whole evaluation will be performed with the same ventilator (ideally the patient's device) using the patient's mask and with the usual ventilator setting.

Measures

At enrolment:

Lung function test Standard questionnaire about the use and tolerability of NIMV at home Measure of NIMV compliance at home Blood gas analysis during wakefulness (during spontaneous breathing - SB - and during NIMV) The breathing pattern during wakefulness (during SB and NIMV)

Polysomnographic evaluation

Full standard assisted polysomnography with simultaneous recordings of Tidal Volume, Leaks, pressure in mask, respiratory rate, instantaneous minute ventilation.

Analysis of sleep data will be performed according to standard criteria (AASM 2007).

Analysis of breathing pattern and patients-ventilator interaction will be made according to previous published methods (Fanfulla, Tuggey, Techsler etc..).

At the end of the each PSG recording, patients will be asked about their humidification and NIMV tolerance as well as the presence of upper airway symptoms (Nava et al).

ELIGIBILITY:
Inclusion Criteria:

* Patients in stable conditions (no acute exacerbations in the 4 weeks before enrolment), well adapted to ventilation and without problems with the ventilation mask.

Exclusion Criteria:

* Patients with acute respiratory failure, recent exacerbations, severe co-morbidities (i.e. hearth failure, recent stroke etc.)
* Recent upper airways surgery.
* Allergic rhinitis, severe nasal stenosis.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-12; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
sleep quality and asynchrony index | 8 hrs

SECONDARY OUTCOMES:
tolerance assessed using an ad-hoc designed scale (1 t0 5 scale), and the effective hours of sleep | 8 hrs

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Fanfulla, MD, Principal Investigator — Fondazione S.Maugeri
Locations (1):
- Fondazione S.Maugeri, Pavia, Pavia, Italy

REFERENCES:
- [Background] Nava S, Cirio S, Fanfulla F, Carlucci A, Navarra A, Negri A, Ceriana P. Comparison of two humidification systems for long-term noninvasive mechanical ventilation. Eur Respir J. 2008 Aug;32(2):460-4. doi: 10.1183/09031936.00000208. PMID 18669787